CLINICAL TRIAL: NCT01450098
Title: Single Dose LY2484595 Tablet Formulations to Determine the Impact of Dose Level, Food, and Ethnicity on the Pharmacokinetics in Healthy Subjects
Brief Title: A Study of LY2484595 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 13697; I1V-MC-EIAJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-10-07; First posted 2011-10-12 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — evacetrapib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A: Fixed Sequence of Meal Conditions (Experimental): LY2484595 (evacetrapib): 200 milligrams (mg) of LY2484595 administered orally, one time only, as an SDSD-PG tablet given with no food. There was a washout of at least 14 days before crossing over and receiving a 200 mg of LY2484595 administered orally, one time only, as a SDSD-PG tablet given with low-fat breakfast. There was another washout period of at least 14 days before crossing over and receiving a 200 mg of LY2484595 administered orally, one time only, as a SDSD-PG tablet given with high-fat breakfast.
  Interventions: Drug: LY2484595 spray-dried solid dispersion-propyl gallate (SDSD-PG)
- Cohort B: Comparison of Randomized Treatments (Experimental): LY2484595 (evacetrapib): 100 mg of LY2484595 administered orally as an RF tablet given with a low-fat breakfast. There was a washout period of at least 14 days before crossing over and receiving 100 mg of LY2484595 administered orally as a SDSD-PG tablet given with a low-fat breakfast. There was another washout of at least 14 days before crossing over and receiving 300 mg of LY2484595 as a SDSD-PG tablet given with a low-fat breakfast.
  Interventions: Drug: LY2484595 Reference Formulation (RF); Drug: LY2484595 spray-dried solid dispersion-propyl gallate (SDSD-PG)

INTERVENTIONS:
Drug: LY2484595 Reference Formulation (RF) — Administered orally
  Other Names: Evacetrapib
  Arms: Cohort B: Comparison of Randomized Treatments
Drug: LY2484595 spray-dried solid dispersion-propyl gallate (SDSD-PG) — Administered orally
  Other Names: Evacetrapib

SUMMARY:
The purpose of this study will be to evaluate the safety of a single dose of LY2484595 and to compare the amount of LY2484595 in the blood of healthy non-Asian subjects, Chinese subjects, and first-generation Japanese subjects after receiving a single oral dose of LY2484595 in a fasted state, after eating a low-fat meal, and after eating a high-fat meal.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination. For Cohort B, a first-generation Japanese subject is defined as one who is Japanese and was born in Japan and whose parents and all grandparents are Japanese and were born in Japan. A first-generation Chinese subject is defined as one who is Chinese and was born in China (mainland or Taiwan) and whose parents and all grandparents are Chinese and were born in China
* Female subjects are not of child-bearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause. Women with an intact uterus are deemed postmenopausal if they are at least age 45, have had cessation of menses for at least 1 year, and have not taken hormones or oral contraceptives (including estrogen or hormone replacement therapy) during the past 12 months
* Have a body mass index (BMI) of 18.5 to 29.0 kilograms per meter squared (kg/m^2), inclusive
* Have clinical laboratory test results within normal reference range for the population or investigator site or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have an acceptable blood pressure (BP) and heart rate at both supine and standing positions as determined by the investigator (systolic BP less than or equal to 140 millimeters of mercury [mmHg], and diastolic BP less than or equal to 90 mmHg). A single, repeat BP measurement may be done at the discretion of the investigator
* Have venous access sufficient to allow blood sampling
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by Eli Lilly and Company (hereafter, Lilly) and the ethical review board (ERB) governing the site

Exclusion Criteria:

* Are currently enrolled in or discontinued within the last 30 days from a clinical trial involving an investigational drug or device or off-label use of a drug or device or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to LY2484595 or related compounds
* Are persons who have previously completed or withdrawn from this study
* Have an abnormality in the 12-lead electrocardiogram (ECG) (including but not limited to a Bazett's corrected QT [QTcB] interval >450 milliseconds (msec) for men and >470 msec for women) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have a history within the last 2 years or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, or neurologic disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Show evidence of significant active neuropsychiatric disease
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Are women with a positive pregnancy test or women who are lactating
* Intend to use and actually use over-the-counter or prescription medication or dietary supplements within 14 days prior to dosing (acetaminophen is permissible on an as-needed basis at less than 3 grams per day for less than 7 days)
* Have donated blood of more than 500 milliliters (mL) within the last month
* Have an average alcohol intake that exceeds 14 units per week, or are unwilling to stop alcohol consumption for 48 hours prior and during the inpatient confinement at the Clinical Research Unit (CRU) (1 unit = 12 ounces [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Use herbal supplements, grapefruit juice, grapefruits, Seville orange juice, Seville oranges, or starfruit within 7 days prior to study dosing
* Smoke more than 10 cigarettes per day currently and are unwilling to abide by the CRU guidelines
* Are unwilling to refrain from daily consumption of real licorice

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri, 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendale, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Fixed Sequence of Meal Conditions: LY2484595: 200 milligrams (mg) of LY2484595 administered orally, one time only, as a spray-dried solid dispersion-propyl gallate (SDSD-PG) tablet given with no food. There was a washout of at least 14 days before crossing over and receiving a 200 mg of LY2484595 administered orally, one time only, as a SDSD-PG tablet given with low-fat breakfast. There was another washout period of at least 14 days before crossing over and receiving a 200 mg of LY2484595 administered orally, one time only, as a SDSD-PG tablet given with high-fat breakfast.
- Cohort B: Comparison of Randomized Treatments: LY2484595: 100 mg of LY2484595 administered orally as reference formulation (RF) tablet given with a low-fat breakfast. There was a washout period of at least 14 days before crossing over and receiving 100 mg of LY2484595 administered orally as a SDSD-PG tablet given with a low-fat breakfast. There was another washout of at least 14 days before crossing over and receiving 300 mg of LY2484595 as a SDSD-PG tablet given with a low-fat breakfast.
Period: Period 1
Arm/Group | Cohort A: Fixed Sequence of Meal Conditions | Cohort B: Comparison of Randomized Treatments
Started | 8 | 31
Received at Least 1 Dose of Study Drug | 8 | 31
Completed | 8 | 31
Not Completed | 0 | 0
Period: Washout Period of at Least 14 Days
Arm/Group | Cohort A: Fixed Sequence of Meal Conditions | Cohort B: Comparison of Randomized Treatments
Started | 8 | 31
Completed | 8 | 31
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Cohort A: Fixed Sequence of Meal Conditions | Cohort B: Comparison of Randomized Treatments
Started | 8 | 31
Received at Least 1 Dose of Study Drug | 8 | 31
Completed | 8 | 31
Not Completed | 0 | 0
Period: Washout of at Least 14 Days
Arm/Group | Cohort A: Fixed Sequence of Meal Conditions | Cohort B: Comparison of Randomized Treatments
Started | 8 | 31
Completed | 8 | 31
Not Completed | 0 | 0
Period: Period 3
Arm/Group | Cohort A: Fixed Sequence of Meal Conditions | Cohort B: Comparison of Randomized Treatments
Started | 8 | 31
Received at Least 1 Dose of Study Drug | 8 | 30
Completed | 8 | 28
Not Completed | 0 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug
Groups:
- Cohort A: Fixed Sequence of Meal Conditions: LY2484595: 200 milligrams (mg) of LY2484595 administered orally, one time only, as an SDSD-PG tablet given with no food. There was a washout of at least 14 days before crossing over and receiving a 200 mg of LY2484595 administered orally, one time only, as an SDSD-PG tablet given with low-fat breakfast. There was another washout period of at least 14 days before crossing over and receiving a 200 mg of LY2484595 administered orally, one time only, as a SDSD-PG tablet given with high-fat breakfast.
- Cohort B: Comparison of Randomized Treatments: LY2484595: 100 mg of LY2484595 administered orally as an RF tablet given with a low-fat breakfast. There was a washout period of at least 14 days before crossing over and receiving 100 mg of LY2484595 administered orally as an SDSD-PG tablet given with a low-fat breakfast. There was another washout of at least 14 days before crossing over and receiving 300 mg of LY2484595 as a SDSD-PG tablet given with a low-fat breakfast.
- Total: Total of all reporting groups
Arm/Group | Cohort A: Fixed Sequence of Meal Conditions | Cohort B: Comparison of Randomized Treatments | Total
Number analyzed (Participants) | 8 | 31 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (6.2) | 37.3 (11.4) | 36.2 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 6 | 6
  Male | 8 | 25 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 6 | 30 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Black or African American | 1 | 3 | 4
  White | 6 | 6 | 12
  Asian (Chinese) | 0 | 10 | 10
  Asian (Japanese) | 0 | 11 | 11
  Multiple | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 31 | 39

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Plasma Concentration Versus Time Curve (AUC) of LY2484595
Description: Area under the concentration-time curve from time zero to infinity is presented.
Time Frame: Predose and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 168 hours postdose
Population: All participants in Cohort A who received at least 1 dose of study drug with evaluable LY2484595 plasma concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours times nanograms per milliliter
Groups:
- LY2484595 200 mg SDSD-PG Fasted: Cohort A: 200 mg of LY2484595 administered orally, one time only as an SDSD-PG tablet given with no food
- LY2484595 200 mg SDSD-PG Low Fat: Cohort A: 200 mg of LY2484595 administered orally, one time only as an SDSD-PG tablet given with a low-fat breakfast
- LY2484595 200 mg SDSD-PG High Fat: Cohort A: 200 mg of LY2484595 administered orally, one time only as an SDSD-PG tablet given with a high-fat breakfast
Arm/Group | LY2484595 200 mg SDSD-PG Fasted | LY2484595 200 mg SDSD-PG Low Fat | LY2484595 200 mg SDSD-PG High Fat
Number analyzed (Participants) | 7 | 8 | 7
hours times nanograms per milliliter | 12200 (29) | 17800 (31) | 17800 (29)

2. Primary Outcome: Pharmacokinetics: Peak Plasma Concentration (Cmax) of LY2484595
Time Frame: Predose and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 168 hours postdose
Population: All participants in Cohort A who received at least 1 dose of study drug with evaluable LY2484595 maximum observed plasma concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | LY2484595 200 mg SDSD-PG Fasted | LY2484595 200 mg SDSD-PG Low Fat | LY2484595 200 mg SDSD-PG High Fat
Number analyzed (Participants) | 8 | 8 | 8
nanograms per milliliter | 828 (51) | 1510 (30) | 1280 (28)

3. Secondary Outcome: Number of Participants With One or More Drug-related Adverse Events (AEs) or Any Serious AEs
Description: Data presented are the number of participants who experienced one or more drug-related AEs or any serious AEs. A summary of serious and other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through completion of study (approximately 2 months)
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: participants
Groups:
- LY2484595 100 mg RF: Cohort B: 100 mg of LY2484595 administered orally one time as an RF tablet with a low-fat breakfast
- LY2484595 100 mg SDSD-PG: Cohort B: 100 mg of LY2484595 administered orally one time as an SDSD-PG tablet with a low-fat breakfast.
- LY2484595 200 mg SDSD-PG: Cohort A: 200 mg of LY2484595 administered orally, one time only as an SDSD-PG tablet given with no food; then, after at least a 14 day washout period, 200 mg of LY2484595 administered orally, one time only, as an SDSD-PG tablet given with a low-fat breakfast; then, after a washout period of at least 14 days, 200 mg of LY2484595 administered orally, one time only, as an SDSD-PG tablet given with a high-fat breakfast
- LY2484595 300 mg SDSD-PG: Cohort B: 300 mg of LY2484595 administered orally one time as an SDSD-PG tablet with a low-fat breakfast.
Arm/Group | LY2484595 100 mg RF | LY2484595 100 mg SDSD-PG | LY2484595 200 mg SDSD-PG | LY2484595 300 mg SDSD-PG
Number analyzed (Participants) | 30 | 30 | 8 | 31
participants | 0 | 0 | 2 | 1

ADVERSE EVENTS:
Arm/Group | LY2484595 100 mg RF | LY2484595 100 mg SDSD-PG | LY2484595 200 mg SDSD-PG | LY2484595 300 mg SDSD-PG
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/8 | 0/31
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 3/8 | 4/31
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2484595 100 mg RF (N=30) | LY2484595 100 mg SDSD-PG (N=30) | LY2484595 200 mg SDSD-PG (N=8) | LY2484595 300 mg SDSD-PG (N=31)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days